CLINICAL TRIAL: NCT06254118
Title: Non-Surgical Treatment of Periodontitis in Menopausal Patients
Brief Title: Treatment of Periodontitis in Menopausal Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hadir F. El-Dessouky (Other)
Responsible Party: Sponsor-Investigator, Hadir F. El-Dessouky, Professor Dr, King Abdulaziz University
Organization: King Abdulaziz University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HElDessouky
Record Dates: First submitted 2024-01-28; First posted 2024-02-12 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Menopausal Patients; Chronic Periodontitis; Omega 3 Fatty Acids
Keywords: Periodontitis, GCF, Osteocalcin.
MeSH Terms: conditions — Chronic Periodontitis; Periodontitis | interventions — Fatty Acids, Unsaturated; Fatty Acids, Omega-3; Olive Oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: an independent researcher not directly involved in the study, utilized a computer generated random number sequence to assign participants to either the control or study group. this randomization was executed before the commencement of the treatment phase.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- group 2 polyunsaturated fatty acids (Experimental): intervention: systemic administration of 1000 mg polyunsaturated fatty acids. to be taken once daily with meals for 12 months
  patients treated by scaling and root planing and oral systemic administration of Omega-3 fatty acids a soft gelatinous capsule containing 1000 mg polyunsaturated fatty acids (PUFAs)
  Interventions: Drug: Polyunsaturated Fatty Acids
- group 1 control (Sham Comparator): control group, patients treated by scaling and root planing and an oral soft gelatinous capsule containing olive oil to be taken once daily with meals for 12 months
  Interventions: Dietary Supplement: olive oil

INTERVENTIONS:
Drug: Polyunsaturated Fatty Acids — 1000mg omega-3 fatty acids taken once daily with meals for 12 months
  Other Names: omega-3 fatty acids
  Arms: group 2 polyunsaturated fatty acids
Dietary Supplement: olive oil — 1000mg olive oil taken once daily with meals for 12 months
  Arms: group 1 control

SUMMARY:
The goal of this clinical trial is to compare the effectiveness of polyunsaturated fatty acids (PUFAs) [omega-3] as an adjunctive treatment to scaling and root planing for menopausal women with periodontitis versus scaling and root alone as a non- surgical treatment .

. The main question it aims to answer is:

• to investigate the effect of systemic administration of Omega-3 fatty acids in addition to SRP on clinical periodontal parameters and GCF levels of osteocalcin and AST in menopausal women.

Participants will given * a soft gelatin capsules containing PUFAs to be consumed directly once daily for 12 months along with non-surgical treatment (group2)

** a soft gelatin capsules containing olive oil to be consumed directly once daily for 12 months along with non-surgical treatment (group1)

Researchers will compare group 1 to group 2 to see if PUFAs has an effect on clinical periodontal parameters and GCF levels of osteocalcin and AST in menopausal women. .

DETAILED DESCRIPTION:
Menopause is typically accompanied by significant systemic and oral manifestations, including hormonal changes and increased susceptibility to periodontal disease, which may involve inflammatory biomarkers like aspartate aminotransferase (AST) and Osteocalcin in gingival crevicular fluid (GCF). The study aims to evaluate the effectiveness of regular inoculation of polyunsaturated fatty acids (PUFAs) as an adjunctive treatment for menopausal women's periodontitis.

Methods: Twenty elderly women with chronic periodontitis were split evenly into two groups by random assignment. Patients in group II (the research group) were given soft gelatin capsules containing PUFAs to be consumed directly once daily for 12 months, as opposed to the group I (the control group), who received soft gelatin capsules containing some olive oil (placebo). Scaling and root planning (SRP) were used to address periodontal disease in all cases.

At baseline, six and twelve months after treatment, clinical indicators and AST and Osteocalcin amounts in the GCF will be noted.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed as; periodontitis patients
* presence of a minimum of 6 teeth in the mouth
* at least 3 periodontal sites with probing pocket depth more or equal to 5mm
* women experiencing menopause for at least a year

Exclusion Criteria:

* women suffering from any systemic disorder that might affect the periodontal tissues such as; Diabetes Mellitus, immune disorders,..
* anemic patients
* smokers
* patients taking NSAIDs, supplements, antibiotics regularly used mouthwashes within the last 3 months
* participants in any other clinical trials

Ages: 45 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2020-01-22 (Actual); Primary Completion 2022-01-22 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
aspartate aminotransferase (AST) in gingival crevicular fluid (GCF). | baseline, 6 months, 12 months
  AST in GCF will be measured in 20 participants, evaluation of AST in the collected GCF. The assessment was done using the VITROS Dry Technology 60 Chemistry System which can provide accurate results using even very small amounts of GCF (~10 µl). The principle behind the test is to evaluate the enzymatic activity of AST to convert the amino group of aspartates where the oxidation process of nicotinamide adenine dinucleotide (NAD) + hydrogen (H) (NADH+). This activity is measured by the Reflectance Spectrophotometry at 340nm wavelength and 37°C. The change in rate assesses the enzymatic activity as per Bergmeyer et al. method.
Osteocalcin in gingival crevicular fluid (GCF). | baseline, 6 months, 12 months
  Osteocalcin in GCF, The evaluation of the level of osteocalcin in the GCF sample, using enzyme-linked immunosorbent assay (ELISA) kits (Ani Biotech Oy, AvioBion, Finland), is the next step in the study. The osteocalcin levels are measured in nanograms per milliliter (ng/mL) when assessed using ELISA kits. The principle applied in the sandwich-type ELISA kit is the presence of a monoclonal osteocalcin which is adsorbed onto the well of the kit and then binds to the osteocalcin (present in the sample). The amount of osteocalcin present was assessed using standard curves based on dilutions and measured at the color intensity of 450nm.

SECONDARY OUTCOMES:
Plaque Index (PI) | baseline, 6 months, 12 months
  The PI was conducted according to O'Leary et al. (1972), this precise index records the presence of supra-gingival plaque on all four tooth surfaces. For this test, the plaque is disclosed using a disclosing tablet. and the stained surfaces around the gingival margins were recorded. the presence or absence of plaque is recorded in a simple chart, the plaque incidence in the oral cavity is expressed as an exact percentage, maximum index is 100%, minimum index is 0%.
Gingival index (GI) | baseline, 6 months, 12 months
  GI was recorded according to Loe and Silness (1963), the gingival index records gingival inflammation in three grades. It is measured on six selected teeth, on facial, lingual, mesial and distal sites. Grades range from 0-3. 0= normal gingiva; no inflammation, no discoloration (erythema), no bleeding. 1= mild inflammation; slight erythema, no bleeding. 2= moderate inflammation; erythema bleeding on probing. (the symptom of bleeding comprises a score of 2). 3= severe inflammation, severe erythema and swelling, tendency to spontaneous bleeding.
Probing pocket depth (PPD) | baseline, 6 months, 12 months
  The examination of PPD was conducted using a UNC-15 periodontal probe (UNC-15, Hu-Friedy, Chicago, IL, USA). PPD was measured at 6 points around each tooth Mesiobuccal (MB), midbuccal (B), Distobuccal (DB), Mesiolingual (ML), midlingual (L), and Distolingual (DL).
  UNC-15 periodontal probe measures 15mm, PPD of 5mm or more were recorded.
Clinical attachment level (CAL) | baseline, 6 months, 12 months
  The examination of CAL was conducted using a UNC-15 periodontal probe (UNC-15, Hu-Friedy, Chicago, IL, USA). CAL was measured at 6 points around each tooth Mesiobuccal (MB), midbuccal (B), Distobuccal (DB), Mesiolingual (ML), midlingual (L), and Distolingual (DL).
  UNC-15 periodontal probe measures 15mm, CAL of 1mm or more were recorded.

CONTACTS AND LOCATIONS:
Overall Officials: ELDESSOUKY, Principal Investigator — King Abdulaziz University
Locations (1):
- King Abdul Aziz University, Jeddah, Mecca Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No
no IPD to be shared

REFERENCES:
- [Derived] Eldessouky HF, Marie M. Nonsurgical Treatment of Periodontitis in Menopausal Patients: A Randomized Control Trial. Biomed Res Int. 2024 Mar 13;2024:6997142. doi: 10.1155/2024/6997142. eCollection 2024. PMID 38510979